CLINICAL TRIAL: NCT01669330
Title: Comparison of Laparoscopic Nissen Versus Anterior Partial Fundoplication ad Modum Watson, A Prospective Randomized Trial
Brief Title: Laparoscopic Nissen Versus Anterior Partial Fundoplication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NW20012011
Record Dates: First submitted 2011-11-22; First posted 2012-08-21 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; Fundoplication; Surgical Procedures
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Fundoplication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total fundoplication (Active Comparator): Procedure: Laparoscopic Nissen fundoplication
  Interventions: Procedure: Nissen fundoplication
- Anterior partial fundoplication (Active Comparator): Procedure: Laparoscopic anterior partial fundoplication
  Interventions: Procedure: Laparoscopic antireflux surgery ad modum Watson

INTERVENTIONS:
Procedure: Nissen fundoplication — Laparoscopic Nissen fundoplication
  Arms: Total fundoplication
Procedure: Laparoscopic antireflux surgery ad modum Watson — Laparoscopic anterior fundoplication
  Arms: Anterior partial fundoplication

SUMMARY:
The most widely used operative technique for gastroesophageal reflux is total fundoplication where the gastric fundus is sutured around the distal esophagus like a wrap. This operation effectively prevents gastroesophageal reflux but gives rise to postoperative symptoms related to over-competence of the gastroesophageal junction. 40% of the operated patients experience increased flatulence and 20% dysphagia. Anterior fundoplication is an alternative technique where the distal esophagus is anchored to the crura of the hiatus esophagi and only a part of the front wall of the esophagus is covered with fundus. An anterior fundoplication is un attempt to create a more physiologic reflux control and less functional problems postoperatively. The aim with this study is to compare the results postoperatively, both short time and long time results.

DETAILED DESCRIPTION:
Aim: To establish if there is a difference in the incidence of postoperative flatulence after the two different operative techniques. The secondary aims are to establish differences in relapse of reflux, incidence of postoperative dysphagia, dyspepsia, quality of life, hospital stay, sick-leave and complications.

Method: All patients operated on for reflux disease in Lund, Malmö,Trollättan and Kalmar are randomised between the two operations. Postoperatively, telephone interview is performed weekly the first two months. One year and ten years postoperatively. The patients are investigated with endoscopy, esophageal manometry, 24 hour pH-monitoring and symptom evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-65 years.
* Good results of PPI treatment (<3 months) resulting in reduced heart burn and acid regurgitations.
* Gastroesophageal reflux disease as evidence by gastroscopy and pH-monitoring.

Exclusion Criteria:

* Previous surgery on the stomach
* Patients with IBS (criteria ROM II)
* Severe disease, for example diabetes mellitus, cardiopulmonary disease or renal disease, that would influence outcome measurement
* Patients with active ulcer disease
* Paraesophageal hernia
* Patient that are incapable to understand the study information (for example mentally disorder, drug abuse)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2001-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Postoperative flatulence? | Postoperative one year
  To establish if there is a difference in the incidence of postoperative flatulence after the two different operative techniques.

SECONDARY OUTCOMES:
Relapse? Complications? Functional problems? | Postoperatively three months, one year and ten years
  To establish differences in relapse of reflux, incidence of postoperative dysphagia, dyspepsia, quality of life, hospital stay, sick-leave and complications.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Djerf, Md, Principal Investigator — Region Skane
Locations (4):
- Sweden (4):
  - Department of Surgery, Kalmar
  - Department of Surgery, Lund
  - Department of Surgery, Malmo
  - Department of Surgery, Trollhättan